CLINICAL TRIAL: NCT03899311
Title: A Protein-sparing Modified Fast for Children and Adolescents With Severe Obesity
Brief Title: A Protein-sparing Modified Fast for Children and Adolescents With Severe Obesity (PSMF)
Acronym: PSMF
Status: Completed | Type: Observational
Sponsor: Ihuoma Eneli (Other)
Responsible Party: Sponsor-Investigator, Ihuoma Eneli, Director, Center for Healthy Weight and Nutrition, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB15-00667
Record Dates: First submitted 2018-01-24; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PSMF cohort: The cohort is instructed to follow a protein-sparing modified fast diet and is given standard health care in the Center for Healthy Weight and Nutrition at Nationwide Children's Hospital.
  Interventions: Other: protein-sparing modified fast diet

INTERVENTIONS:
Other: protein-sparing modified fast diet — a PSMF diet follow the usual care format in the Center
  Other Names: The PSMF diet

SUMMARY:
This is a 12 month prospective observational cohort study of the outpatient protein-sparing modified fast diet for children with severe obesity and serious comorbid condition(s). The study will enroll 30 Center for Healthy Weight and Nutrition patients aged 11-19 years who have been placed on a protein sparing modified fast as part of their treatment plan. The study-specific procedures consist of questionnaires/interviews on diet and PA behaviors, adherence and self-efficacy measures, data abstraction from the chart and tracking of activity using a Fitbit.

DETAILED DESCRIPTION:
Aggressive dietary interventions may provide an accessible treatment option for children and adolescents with severe obesity who are not successful with traditional lifestyle behavioral interventions or do not want or qualify for weight loss surgery. One such intensive dietary option is the protein sparing modified fast (PSMF). The PSMF involves minimal carbohydrate intake to induce ketosis, while maintaining adequate or high protein intake to minimize catabolism. The PSMF, under medical supervision, can be an effective and safe intervention for children and adolescents, yet the PSMF diet is not regularly used in the treatment of pediatric severe obesity. This pilot study will employ a prospective cohort study design. Thirty children, 11-19 years-old, with severe obesity, who have been prescribed the rPSMF as part of their treatment in a tertiary care pediatric weight management clinic (PWMC), will be recruited along with their attending parent to participate in the study. The primary aim of the study is to evaluate the acceptability of the rPSMF as assessed by adherence, satisfaction with the intervention, and participation rate using quantitative and qualitative methods. The secondary aim is to investigate the effectiveness of the rPSMF on improving a) anthropometric measures (weight, body mass index [BMI] and BMI z-score); b) metabolic measures (lipid profile, glycosylated hemoglobin, liver function tests); and c) quality of life. Results of this study will provide guidance for the standardization of a pediatric rPSMF protocol in a clinic setting, delineate which factors improve or hinder adherence and weight loss and provide preliminary data for a multicenter randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Children Age 11-19 years old
* Must be severely obese (BMI greater than or equal to 120% of the 95th percentile for their age and sex, or a BMI of 35 or greater)
* Must have at least one severe comorbidity
* Tanner Stage III, IV, V

Exclusion Criteria:

* non-English speaking
* Patients without adequate social/psychological capacity, as evidenced by unavailability to recourses, or family is unable to provide support.

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents seen by Center for Healthy Weight and Nutrition at Nationwide Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
The acceptability of PSMF diet in a tertiary weight management clinic | Baseline
  The percentage of patients and families recruited over all approached eligible patients, during the recruitment period
The acceptability of PSMF diet in a tertiary weight management clinic | 12 months
  Adherence to the diet tracked by clinical dietitian's notes

SECONDARY OUTCOMES:
Change of body weight between baseline and 12 months among subjects on PSMF | Baseline and 12 months
  Body weight in kilograms
Change of Body Mass Index (BMI) between baseline and 12 months among subjects on PSMF | Baseline and 12 months
  BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Ihuoma Eneli, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watowicz RP, Tindall AL, Hummel JC, Eneli IU. The Protein-Sparing Modified Fast for Adolescents With Severe Obesity. Childhood Obesity and Nutrition 7(5): 233-241, 2015.
- [Derived] Eneli IU, Watowicz RP, Xu J, Tindall A, Walston M, Tanner K, Worthington J, Pratt KJ. Rationale and design of a pilot study to evaluate the acceptability and effectiveness of a revised protein sparing modified fast (rPSMF) for severe obesity in a pediatric tertiary care weight management clinic. Contemp Clin Trials Commun. 2019 May 27;15:100388. doi: 10.1016/j.conctc.2019.100388. eCollection 2019 Sep. PMID 31431932